CLINICAL TRIAL: NCT02042339
Title: Hyperbaric Oxygenation (HBO) in Chronic Diabetic Leg Ulcer.
Brief Title: Hyperbaric Oxygenation in Diabetic Ulcer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-265ex11/12; 2012-001436-57 (EudraCT Number)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus
Keywords: Hyperbaric Oxygen; Diabetic ulcer; Wound healing; 3-D life-viz- system; Indocyanine green video angiography; Transcutaneous oxygen pressure; Endothelial progenitor cells
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen (Experimental): Problem-wound schedule: 2.4 atmospheres, 100% oxygen for 90 minutes, two 10 - minute breaks (patients breathing pressurized air from the chamber atmosphere)
  Interventions: Drug: Hyperbaric oxygen
- Sham Hyperbaric oxygen (Placebo Comparator): The patients will be transferred into the chamber like the treatment group. Instead of 100% oxygen they will breathe normal air through the tight fitting masks, at an ambient pressure of 1.1 bar. During the two 10 - minute breaks patients will breathe pressurized air from the chamber atmosphere.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — The treatment will be applied in a large walk-in drive-in hyperbaric chamber. Depending on their general condition, the patients will sit in comfortable chairs or remain in their own wheelchair or bed in relaxed position. They will be accompanied by a medical attendant or by a hyperbaric physician if necessary due to their general condition. Oxygen 100% will be distributed over a tight fitting oxygen-mask connected to the overboard-dumping system. The treatment will be administered according to the so-called problem-wound schedule once a day for six consecutive weeks. On weekends and on public holidays the patients will be off therapy.
  Other Names: HBO; Hyperbaric oxygenation

SUMMARY:
Hyperbaric oxygenation (HBO) involves breathing of 100% oxygen under elevated ambient pressure. In correlation to the pressure level oxygen dissolves in the plasma resulting in an increase of total oxygen in the body. The elevated tissue levels of oxygen may persist for hours, instigating healing processes in wounds caused by disturbances in of perfusion in small vessels, a condition often found in patient with diabetes.

We plan a prospective, double-blind randomized clinical study in 80 patients with chronic diabetic ulcer. All will have optimum treatment of diabetes. The HBO group will be given HBO at 2.4 bar, 90 min., 30 sessions, controls will have sham HBO. Routine wound care will be identical in both groups. Before, during and after treatment (3, 6 and 12 months), a number of monitoring and imaging procedures will be done, cells in the bloodstream indicating improved healing will be determined.

Hypothesis: HBO will instigate the healing process in the majority of patients with chronic diabetic leg ulcer, provided the patency of the large vessels is given.

DETAILED DESCRIPTION:
We plan a prospective, double-blind randomized clinical study (phase III) in 80 patients with diabetes mellitus. All of them will receive the optimum metabolic treatment for their underlying disease. The treatment group will be administered HBO according to the problem wound schedule, the controls will have sham treatment in the hyperbaric chamber. Routine wound care (dressings, physiotherapy, antibiotics if necessary) will be identical in both groups and according to its clinical needs.

Before treatment, indocyanine green videoangiography (ICG), transcutaneous (partial) oxygen pressure (TcPO2) and LifeViz 3D (three-dimensional medical imaging and reconstruction) documentation will be done and endothelial progenitor cells (EPC) as well as markers of bone metabolism will be determined in all patients.

The measurements will be repeated according to the schedule during the treatment period and at controls after 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Age between 18 and 80 years
* Chronic foot ulcer (up to Wagner scale III)
* Patency of large vessels tributary to region of wound
* Good outpatient diabetes management as verified by a specialized centre (HbA1c<8.5%; IFCC: 69mmol/mol).

Exclusion Criteria:

* Clinically relevant obstruction of large vessels tributary to region of wound
* Non-adherence to diabetes therapy
* Pregnancy
* Reactive airway disease
* Radiographic evidence of pulmonary blebs or bullae
* Untreated pneumothorax
* History of seizures except childhood febrile seizures
* Cardiovascular instability
* Mechanical ventilator support
* Treatment with Bleomycin or Anthracyclin in history
* Unable to perform the Valsalva-procedure
* Participation as a subject in any other medical or biomedical research project; if previously involved as a subject, sufficient time must have elapsed to permit "wash out" of any investigational agent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
ICG (indocyanine green) video angiography | Weeks 1-3, 6; Months 3, 6, 12
  Change in ICG-adsorption measured by ICG video angiography from baseline to week/month xxx

SECONDARY OUTCOMES:
High performance 3D LifeViz™ system | Week 1-6; Months 3, 6, 12
  Change of size/configuration of wound from baseline to week/month xxx

OTHER OUTCOMES:
Endothelial progenitor cells | Weeks 1-6, Months 3,6,12
  Modulation of number

CONTACTS AND LOCATIONS:
Overall Officials: Freyja M Smolle-Juettner, M.D., Principal Investigator — Medical University of Graz
Locations (1):
- Division of Thoracic and Hyperbaric Surgery, Graz, Styria, Austria

REFERENCES:
- [Result] O'Reilly D, Pasricha A, Campbell K, Burke N, Assasi N, Bowen JM, Tarride JE, Goeree R. Hyperbaric oxygen therapy for diabetic ulcers: systematic review and meta-analysis. Int J Technol Assess Health Care. 2013 Jul;29(3):269-81. doi: 10.1017/S0266462313000263. PMID 23863187
- [Result] Londahl M. Hyperbaric oxygen therapy as adjunctive treatment of diabetic foot ulcers. Med Clin North Am. 2013 Sep;97(5):957-80. doi: 10.1016/j.mcna.2013.04.004. Epub 2013 Jul 6. PMID 23992903
- [Result] Kranke P, Bennett MH, Martyn-St James M, Schnabel A, Debus SE. Hyperbaric oxygen therapy for chronic wounds. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD004123. doi: 10.1002/14651858.CD004123.pub3. PMID 22513920
- See also: The Division of Thoracic and Hyperbaric Surgery is part of the Medical University Graz — http://www.medunigraz.at/